CLINICAL TRIAL: NCT00669370
Title: Biweekly Docetaxel (Taxotere®)in Combination With Capecitabine (Xeloda®)as First-Line Treatment in Patients With Advanced Gastric Cancer
Brief Title: Biweekly Docetaxel in Combination With Capecitabine as First-Line Treatment in Patients With Advanced Gastric Cancer
Acronym: GAST-TaxXel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Raija Ristamäki, Department of Oncology and Radiotherapy, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002484-87; EudraCT no 2005-002484-87
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Stomach Neoplasms
Keywords: advanced gastric cancer; adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel and capecitabine — biweekly docetaxel iv (50 mg/m2) on day 1 and 15 and capecitabine po 1250 mg/m2 x 2/day days 1-7 and 15-21, treatment cycle consisting of 21 days
  Other Names: Taxotere; Xeloda

SUMMARY:
To determine the quality of life in patients with gastric cancer who receive combination treatment with docetaxel and capecitabine. Secondary endpoints are time to progression, overall response rate and overall survival.

Study treatment will continue until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
GAST-TaxXel is an open, phase II, single arm, non-randomized, Finnish multicenter trial. At least 50 subjects will be enrolled.

Primary endpoint:

To determine the quality of life (EORTC QLQ-C30 and QLQ-STO22) in patients with gastric cancer who receive combination treatment with Taxotere and Xeloda.

Secondary endpoint:

To evaluate time to progression (TTP), overall response rate (ORR) and overall survival (OS).

Quality of life: to evaluate that QOL does not deteriorate from baseline. Quality of life is measured using EORTC QLQ-C30 and QLQ-STO22 with physical functioning score as the primary variable.

Efficacy: time to progression, overall response rate, overall survival Time to progression is defined as time elapsed from inclusion to first documented progression or death whatever the reason. Overall response rate is assessed according to the RECIST criteria. Overall survival is defined as time elapsed from inclusion to death.

Safety: clinical and laboratory toxicities or symptomatology will be graded according to NCI-CTC criteria.

Statistical considerations:

The primary variable, physical functioning score measured by the EORTC QLQ-C30 and QLQ-STO22 instrument, will be analyzed using a paired t-test (change from baseline after two treatment cycles). A 95% confidence interval will also be calculated for the primary variable. Median TTP and OS will be estimated using the Kaplan-Meier method. The ORR will be summarized. Safety variables will be summarized descriptively.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed advanced, inoperable gastric adenocarcinoma
* age ≥18 years
* WHO performance status ≤ 2
* Stage IV
* Measurable (according to RECIST criteria) or evaluable lesion
* No previous chemotherapy, except adjuvant chemotherapy ≥ 6 months ago
* Adequate hematological function (neutrophils ≥ 1.5 x 109/l and platelets ≥ 100 x 109/l, Hb ≥ 100 g/l (after transfusion when needed)
* Adequate renal function (serum creatinine ≤ 1.25 x upper normal limit)
* Adequate liver function (total serum bilirubin ≤ 1.25 x upper normal limit or ALAT ≤ 3 x upper normal limit; in case of liver metastasis: total serum bilirubin ≤ 1.5 x upper normal limit, ALAT ≤ 5 x upper normal limit)
* AFOS ≤ 2.5 x upper normal limit (unless bone metastases)
* Consent form signed and dated before inclusion
* Able to comply with the scheduled follow-up and with the management of toxicities.

Exclusion Criteria:

* Pregnant or lactating women (or potentially fertile women not using adequate contraception)
* Presence of CNS metastases
* Unresolved bowel obstruction or subobstruction
* Chronic diarrhea
* Clinically significant malabsorption syndrome
* Inability to swallow tablets
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Concurrent severe and/or uncontrolled co-morbid medical condition such as uncontrolled infection, hypertension, ischemic heart disease, myocardial infarction within previous 6 months, congestive heart failure
* History of previous or concurrent malignancy within the previous 5 years except curatively treated carcinoma in situ of the uterine cervix or basal cell carcinoma of the skin
* History of prior serious allergic reactions such as anaphylactic shock.
* Peripheral neuropathy ≥ grade 2, unless related to mechanical etiology
* Concurrent use of corticosteroids unless chronic treatment (i.e. initiated > 6 months prior to study entry) at low doses (≥ 20 mg methylprednisolone or equivalent)
* History of allergy to drugs containing the excipient TWEEN 80® and/ or 5- fluorouracil.
* Lack of physical integrity of the upper gastrointestinal tract.
* Concomitant administration of any other experimental drug under investigation: concurrent treatment with any other anti-cancer therapy.
* Major surgery within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* Patients who cannot be regularly followed up for psychological, social, family or geographic reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To determine the quality of life (EORTC QLQ-C30 and QLQ-STO22) | at baseline and on day 1 at every cycle, at the end of study and every 8 week until progress

SECONDARY OUTCOMES:
To evaluate time to progression (TTP), overall response rate (ORR) and overall survival (OS). | every 3 cycles, at the end of study and every 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Raija Ristamäki, MD, PhD, Principal Investigator — Department of Oncology and Radiotherapy, Turku University Hospital
Locations (6):
- Finland (6):
  - Kuopio University Hospital, Kuopio
  - Oulu Univerity Hospital, Oulu
  - Satakunta District Hospital, Pori
  - University of Tampere, Tampere
  - Department of Oncology and Radiotherapy, turku University Hospital, Turku
  - Vaasa Distric Hospital, Vaasa

REFERENCES:
- [Derived] Korkeila EA, Salminen T, Kallio R, Mikkola M, Auvinen P, Pyrhonen S, Ristamaki R. Quality of life with biweekly docetaxel and capecitabine in advanced gastro-oesophageal cancer. Support Care Cancer. 2017 Sep;25(9):2771-2777. doi: 10.1007/s00520-017-3689-5. Epub 2017 Apr 20. PMID 28424889